CLINICAL TRIAL: NCT06985641
Title: Home-Based Community Health Worker Support for Mental Health Among People Living With HIV in South Africa: A Hybrid Effectiveness Implementation Trial
Brief Title: Khanya Ekhaya: A Home-Based Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: Medical Research Council, South Africa (Other); Fogarty International Center of the National Institute of Health (NIH); Curtin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC017-8/2024; 1R21TW012347-01A1 (NIH)
Record Dates: First submitted 2025-04-29; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: HIV; HIV Antiretroviral Therapy (ART) Adherence; Mental Health; Substance Use Disorders; Stigma; Community Health Workers; Training; Global Health; Mental Health Recovery; Substance Use Recovery
Keywords: Community Health Workers; Health Personnel; Global Health; Substance Use Recovery; Mental Health Recovery; HIV; Health Care Seeking Behavior; Treatment Adherence and Compliance; Attitude of Health Personnel; Substance Use Stigma; Mental health Stigma; Substance Use Disorders
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders; Social Stigma; Patient Acceptance of Health Care; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: The intervention will be delivered in Aim 3 (clinical trial). This study uses a parallel design. Two existing teams of healthcare workers will be randomized 1:1 at the team level to receive the Khanya-Ekhaya training or to continue their patient care as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Treatment As Usual (No Intervention): This site will receive enhanced treatment as usual (ETAU)-a one-day training for all CHWs on mental health screening, psychoeducation on mental health in HIV and impact on HIV care outcomes, and available referral pathways, and encouraged to use these skills during their home visits.
- Khanya-Ekhaya (Experimental): The Khanya Ekhaya intervention includes an integration of several evidence-based treatment components, including motivational interviewing (MI), problem solving therapy (PST), and behavioral activation (BA), previously tested and adapted for this context in clinic settings, as well as cognitive-behavioral and mindfulness strategies that target rumination and negative thinking patterns. Aims 1-2 will inform Khanya-Ekhaya adaptation, including intervention length, but it is likely to include 3-6 sessions of CHW home visits based on formative work with ongoing supervision and support for CHWs.
  Interventions: Behavioral: Khanya-Ekhaya

INTERVENTIONS:
Behavioral: Khanya-Ekhaya — The Khanya Ekhaya intervention includes an integration of several evidence-based treatment components, including motivational interviewing (MI), problem solving therapy (PST), and behavioral activation (BA), previously tested and adapted for this context in clinic settings, as well as cognitive-behavioral and mindfulness strategies that target rumination and negative thinking patterns. Aims 1-2 will inform Khanya-Ekhaya adaptation, including intervention length, but it is likely to include 3-6 sessions of CHW home visits based on formative work with ongoing supervision and support for CHWs.
  Arms: Khanya-Ekhaya

SUMMARY:
Mental health conditions, such as depression, anxiety, and harmful alcohol use are prevalent among people with chronic diseases, including HIV, and contribute to poor engagement in care. There is a need to address untreated mental health problems. Community health workers (CHWs) are frontline workers who play a central role in supporting vulnerable individuals to stay in care, including seeking people living with HIV who are newly initiating antiretroviral therapy (ART) or re-initiating after a period of care disengagement. CHW-delivered interventions are promising for improving engagement and retention in care. Yet, these programs rarely address mental health -a significant barrier to chronic disease care engagement and treatment. An approach that moves beyond providing care in the clinic setting is needed. Community-delivered home-based mental health care has been shown to be feasible and acceptable and shows promise for integration into broader community health care services for people with chronic conditions, such as HIV.

DETAILED DESCRIPTION:
The overall aim of this 3-phase study (the third phase being the clinical trial) is to develop a feasible mental health intervention for CHW delivery during home-based care for people with chronic conditions, including HIV. Investigators will use an existing cadre of CHWs conducting home visits, highlighting the potential for sustainability.

Aim 1: To explore barriers and facilitators to implementing a home-based, CHW-delivered intervention for mental health concerns (depression, anxiety, harmful alcohol use) "Khanya-Ekhaya". Guided by the Consolidated Framework for Implementation Research (CFIR), investigators will accomplish this aim by conducting individual semi-structured interviews with CHWs and other key stakeholders, including CHW supervisors, policymakers, and organizational leaders and patients with mental health problems. Key domains of the interviews include: (a) appropriateness of providing integrated home-based care for mental health among people newly initiating or re-initiating HIV services after ≥3 months; (b) barriers and facilitators to implementing a CHW-delivered intervention for mental health and HIV care engagement in patients' homes, including how to promote feasibility within CHWs' existing roles; (c) training and supervision needs of CHWs, including how to manage risk and support referrals; and (d) adapting existing evidence-based intervention components developed by the research team (problem solving, motivational interviewing, behavioral activation, mindfulness) for CHW home-delivery.

Aim 2: To adapt with patients and CHWs a home-based, intervention to improve mental health symptoms and HIV outcomes "Khanya-Ekhaya". Investigators will adapt a home-based CHW intervention ("Khanya-Ekhaya" or "Khanya at home") to address mental health symptoms and improve HIV care engagement based on our formative clinic-based work and training CHWs in reducing mental health stigma refined based on Aim 1 feedback. Adapting the intervention components from clinic-based delivery to CHW home-based delivery will be heavily guided by qualitative analysis in Aim 1.

Aim 3 (Clinical Trial). To evaluate the implementation and preliminary effectiveness of a home-based CHW intervention "Khanya-Ekhaya" to reduce mental health symptoms and improve engagement in HIV care. In a pilot Type 1 hybrid effectiveness-implementation trial, investigators will evaluate the effectiveness and implementation of the Khanya-Ekhaya home-delivered CHW intervention. This trial will demonstrate successful training of CHWs, reaching patients of interest, and collecting primary outcomes to inform future work.

ELIGIBILITY:
Inclusion Criteria:

CHWs:

* at least 18 years old
* must conduct home visits for people with HIV newly initiating or re-initiating ART at the approved clinic site

PATIENTS:

* at least 18 years old
* seen by a CHW after newly initiating or re-initiating ART in the past three months
* screen positive for depressive symptoms or harmful alcohol use

Exclusion Criteria:

CHWs:

-Unable or unwilling to complete informed consent and study procedures in English, isiXhosa, or Afrikaans

PATIENTS:

-Unable or unwilling to complete informed consent and study procedures in English, isiXhosa, or Afrikaans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Khanya Ekhaya | 3-month follow-up assessment
  Feasibility is defined as the suitability and practicability of Khanya Ekhaya intervention and implementation strategies. This will be measured via (1) 14-item feasibility subscale of Applied Mental Health Research (AMHR) group implementation measure (scored 0-3).
Acceptability of Khanya Ekhaya | 3-month follow-up assessment
  Acceptability of Khanya Ekhaya is defined as satisfaction, relevance, usefulness of CHW intervention and implementation strategies, measured via a 15-item acceptability subscale of AMHR implementation measure (scored 0-3).
HIV Care Engagement | 3-month follow-up assessment
  HIV care engagement is defined as the proportion of people with HIV (patients) receiving care after first CHW visit and monthly appointment attendance. Receipt of HIV care services will be assessed via medical records, including appointment attendance

SECONDARY OUTCOMES:
Fidelity of CHW delivery | 3-month follow-up assessment
  Fidelity monitoring of delivery of intervention components and competence will be assessed using the (ENhancing Assessment of Common Therapeutic factors) ENACT scale for the Khanya-Ekhaya group.
Fidelity of ETAU | 3-month follow-up assessment
  Fidelity to ETAU will be assessed via documentation of screening and referrals.
Mental health - depressive symptoms | 3-month follow-up assessment
  Mental health symptoms will be assessed among patients using routine mental health screening data extracted from patients' medical records using the Patient Health Questionnaire-2 (PHQ-2) to measure depressive symptoms
Mental health - alcohol use | 3-month follow-up assessment
  Mental health symptoms will be assessed among patients using routine mental health screening data extracted from patients' medical records using the Alcohol Use Disorders Identification Test (AUDIT-C) to measure alcohol use.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica F Magidson, PhD, Principal Investigator — University of Maryland, College Park; Tara Carney, PhD, Principal Investigator — Medical Research Council, South Africa; Bronwyn Myers, PhD, Principal Investigator — Curtin University; South African Medical Research Council
Locations (1):
- South African Medical Research Council - Delft Office, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Investigators will provide de-identified transcripts, codebooks, and quantitative data from this project to interested individuals (with appropriate training and approvals) upon completion of each study aim. These data will be provided in digital format with clear labels for all variables. Data will be released directly by the investigators providing evidence of their institution's IRB approval for planned analyses of the data. Our team will be available to address queries.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available following completion of each study aim (i.e., after publication of the main outcome paper).
Access Criteria: Data will be released directly by the investigators to interested individuals providing evidence of their institution's IRB approval for planned analyses of the data.